CLINICAL TRIAL: NCT02142166
Title: Die Rolle Der Biomarker in Serum, Liquor Und Parenchym im Rahmen Der Aneurysmatischen Subarachnoidalblutung: Verlauf Und Korrelation zu Therapie Und Outcome - bioSAB -
Brief Title: The Role of Biomarker in Serum, Cerebrospinal Fluid and Parenchyma in the Context of Aneurysmal Subarachnoid Hemorrhage.
Acronym: bioSAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Walid Albanna, Priv.-Doz. Dr. med. Walid Albanna, RWTH Aachen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTC-A 14-004
Record Dates: First submitted 2014-04-30; First posted 2014-05-20 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: aneurysmal subarachnoid hemorrhage (ASH); biomarker
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAB analysis (Experimental): Patients with acute aneurysmal SAH, confirmed by CT or MRI, or lumbar puncture
  Daily (21 days) analysis of Biomarker in serum, in liquor and in micro-dialysate
  Interventions: Procedure: Biomarker in serum, liquor, micro-dialysate
- Control (Experimental): Patients who undergo a lumbar puncture for myelography as part of the investigation of a cervical or lumbar foraminal stenosis without cranial or myeläre pathology -or- Patients who receive perioperative prophylactic lumbar drainage without cranial or myeläre pathology
  Single analysis of Biomarker in serum and liquor
  Interventions: Procedure: Biomarker in serum and in liquor

INTERVENTIONS:
Procedure: Biomarker in serum, liquor, micro-dialysate — Daily (21 days) analysis of biomarker in serum, in liquor and in micro-dialysate
  Arms: SAB analysis
Procedure: Biomarker in serum and in liquor — Single analysis of biomarker in serum and liquor
  Arms: Control

SUMMARY:
The aim of this study is to improve the usability of biomarkers for the timely prediction of new complications following a cerebral hemorrhage, especially in combination with invasive, functional and local measurements for patients with aneurysmal subarachnoid hemorrhage (SAH). Based on analyzed biomarker profiles the chosen therapy efforts are assessed in their immediate and longer-term effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* male or female, age ≥ 18 years
* signed consent for participation in the study
* signed consent for further analysis of the samples collected during the clinical routine
* in-patients

Exclusion Criteria:

* female or male patient <18 years
* pregnancy, lactation
* lack of signed informed consent for participation in the study
* lack of signed consent for the further analysis of the samples collected during the clinical routine
* taking a study drug within the last thirty days
* Simultaneous participation in another clinical trial (except participation as control group)
* persons who are in a dependent relationship or employment with the sponsor or investigator
* persons housed for a judicial or administrative order in an institution

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Biomarker in serum, cerebrospinal fluid and parenchyma after aneurysmal SAH | Each participant will be followed at hospital stay for an expected average of 3 weeks. The outcome measure will be assessed after 24 month.
  Temporal development of alternative biomarkers in serum, cerebrospinal fluid and parenchyma after aneurysmal SAH, and their response as influenced by the treatment path.

SECONDARY OUTCOMES:
Clinical outcome | Each participant will be followed at hospital stay for an expected average of 3 weeks. The outcome measure will be assessed after 24 month
  Clinical outcome of patients depending on treatment algorithm and observed development of alternative biomarkers
Image morphological outcome | Each participant will be followed at hospital stay for an expected average of 3 weeks. The outcome measure will be assessed after 24 month
  Image morphological outcome of patients depending on treatment algorithm and observed development of alternative biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Walid Albanna, Priv.-Doz. Dr. med., Principal Investigator — Department of Neurosurgery, University Hospital RWTH Aachen
Locations (1):
- Department of Neurosurgery, University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Neumaier F, Stoppe C, Stoykova A, Weiss M, Veldeman M, Hollig A, Hamou HA, Temel Y, Conzen C, Schmidt TP, Dogan R, Wiesmann M, Clusmann H, Schubert GA, Haeren RHL, Albanna W. Elevated concentrations of macrophage migration inhibitory factor in serum and cerebral microdialysate are associated with delayed cerebral ischemia after aneurysmal subarachnoid hemorrhage. Front Neurol. 2023 Jan 13;13:1066724. doi: 10.3389/fneur.2022.1066724. eCollection 2022. PMID 36712451
- [Derived] Veldeman M, Weiss M, Albanna W, Nikoubashman O, Schulze-Steinen H, Clusmann H, Hoellig A, Schubert GA. Incremental Versus Immediate Induction of Hypertension in the Treatment of Delayed Cerebral Ischemia After Subarachnoid Hemorrhage. Neurocrit Care. 2022 Jun;36(3):702-714. doi: 10.1007/s12028-022-01466-7. Epub 2022 Mar 8. PMID 35260962
- [Derived] Conzen C, Weiss M, Albanna W, Seyfried K, Schmidt TP, Nikoubashman O, Stoppe C, Clusmann H, Schubert GA. Baseline characteristics and outcome for aneurysmal versus non-aneurysmal subarachnoid hemorrhage: a prospective cohort study. Neurosurg Rev. 2022 Apr;45(2):1413-1420. doi: 10.1007/s10143-021-01650-x. Epub 2021 Oct 4. PMID 34604940
- [Derived] Veldeman M, Weiss M, Simon TP, Hoellig A, Clusmann H, Albanna W. Body mass index and leptin levels in serum and cerebrospinal fluid in relation to delayed cerebral ischemia and outcome after aneurysmal subarachnoid hemorrhage. Neurosurg Rev. 2021 Dec;44(6):3547-3556. doi: 10.1007/s10143-021-01541-1. Epub 2021 Apr 17. PMID 33866464
- [Derived] Veldeman M, Lepore D, Hollig A, Clusmann H, Stoppe C, Schubert GA, Albanna W. Procalcitonin in the context of delayed cerebral ischemia after aneurysmal subarachnoid hemorrhage. J Neurosurg. 2020 Sep 4;135(1):29-37. doi: 10.3171/2020.5.JNS201337. Print 2021 Jul 1. PMID 32886914